CLINICAL TRIAL: NCT03192072
Title: Evaluation of a Rapid Diagnostic Test for the Categorization of Acute Respiratory Illness
Brief Title: A Rapid Test for Acute Respiratory Illness
Acronym: Radical
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Antibacterial Resistance Leadership Group (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00082317; Pro00082322 (Other: Duke UMC)
Record Dates: First submitted 2017-06-16; First posted 2017-06-19 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Respiratory Tract Infection Acute; Transcriptome; Virus Disease; Bacterial Infections
MeSH Terms: conditions — Virus Diseases; Bacterial Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Samples will include blood, urine, nasopharyngeal and throat swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Subjects with Acute Respiratory Illness: Patients with acute respiratory illness identified in the Emergency Department
  Interventions: Diagnostic Test: Host Gene Expression

INTERVENTIONS:
Diagnostic Test: Host Gene Expression — comparison to retrospective clinical adjudication
  Other Names: Adjudication

SUMMARY:
The primary purpose of this study is to support the development of a host response test for acute respiratory illness to identify bacterial, viral or NB/NV etiologies as compared to a clinical adjudication reference standard.

Secondary objectives include:

1. Evaluate the effect of age on the performance of the HR-ARI test
2. Evaluate the effect of race/ethnicity on the performance of the HR-ARI test
3. Evaluate the effect of geography on the performance of the HR-ARI test

DETAILED DESCRIPTION:
The primary purpose of this study is to support the development of a host response test for acute respiratory illness to identify bacterial, viral or NB/NV etiologies as compared to a clinical adjudication reference standard.

Secondary objectives include:

1. Evaluate the effect of age on the performance of the HR-ARI test
2. Evaluate the effect of race/ethnicity on the performance of the HR-ARI test
3. Evaluate the effect of geography on the performance of the HR-ARI test

Subjects will be identified in the Emergency Department of participating hospitals. Samples including nasopharyngeal swab, throat swab, blood, and urine will be obtained.

A case report form for each subject will be completed to include information regarding clinical characteristics, signs and symptoms of infection, presence of complications, and patient outcome. Baseline characteristics including preexisting conditions. Survival data will also be collected for each subject.

Samples collected will be used to characterize the patient's illness as either infectious or not, and if infectious, either bacterial or viral. Samples will also be used to measure changes in gene expression, referred to as the Host Response-Acute Respiratory Illness (HR-ARI) test.

The result of this test will be made in comparison to a retrospective review of the subject's clinical information. Results will not be used for any interventions and will not be released to subjects or their providers.

Because the study procedure includes only sample and data collection, the risks will be minimal and no different than encountered during routine clinical care.

The study was re-assessed in 2020 and applicable updates were made to the record.

ELIGIBILITY:
Inclusion Criteria:

A. Age 24 months or older

B. Acute respiratory illness of less than 28 days in duration.

C. Acute respiratory illness will be defined by at least two qualifying symptoms OR one qualifying symptom and at least 1 qualifying vital sign abnormality:

* Qualifying symptoms:Headache, rhinorrhea, nasal congestion, sneezing, sore throat, itchy or watery eyes, conjunctivitis, cough, shortness of breath, sputum production, chest pain, wheezing
* Qualifying Vital Signs: Age greater than or equal to 2 and less than 6:Tachycardia (HR greater than or equal to 110), Tachynpnea (RR greater than or equal to 20),Temperature greater than or equal to 38.5 degrees Celsius or less than or equal to 36 degrees Celsius. Age greater than or equal to 6: Tachycardia(HR greater than or equal to 90), Tachynpnea (RR greater than or equal to 20), Temperature greater than or equal to 38.5 degrees Celsius or less than or equal to 36 degrees Celsius.

D. Ability of the subject or legally authorized representative/parent to understand study procedures, and willing and able to comply with all required.

Exclusion Criteria:

A. Known or suspected infection at any other anatomic site requiring antibacterial therapy.

B. Any specific condition that in the judgment of the referring provider or the site investigator precludes participation because it could affect subject safety or ability of subject to participate in this trial.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Up to 750 subjects may be enrolled at a minimum of 3 study sites from geographically diverse locations across the US. Subjects will be approached based on symptoms upon presentation to the health care facility's ED. In addition to these subjects, data from 450 previously enrolled subjects will be used. All demographic groups will have access to enrollment because anyone with acute respiratory infection (ARI) will be approached. Foreign language speaking subjects may be enrolled following review and approval of the appropriate consent process and documents by the reviewing IRB.
Sampling Method: Probability Sample
Enrollment: 783 (Actual)
Dates: Start 2017-07-17 (Actual); Primary Completion 2019-09-06 (Actual); Study Completion 2019-12-19 (Actual)

PRIMARY OUTCOMES:
Positive predictive value with reference standard (PPV) | Day 1
  Number of assay positives that agree with the reference standard / [Number of assay positives that agree with the reference standard + Number of assay positives that disagree with the reference standard]
Negative predictive value with the reference standard (NPV) | Day 1
  Number of assay negatives that agree with the reference standard / [number of assay negatives that agree with the reference standard + number of assay negatives that disagree with the reference standard]

SECONDARY OUTCOMES:
Overall agreement with the reference standard (OA) | Day 1
  Number of samples that agree with the reference standard / all samples tested

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Woods, MD, MPH, Principal Investigator — Duke University
Locations (10):
- United States (10):
  - The University of California- Davis, Davis, California
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Newton-Wellesley Hospital, Newton, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Rhode Island/Lifespan, Providence, Rhode Island
  - The University of Texas- Houston, Houston, Texas
  - University of Utah Medical Center, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No